CLINICAL TRIAL: NCT03111901
Title: Low-dose Interleukin-2 and Pembrolizumab Among Patients With Metastatic Melanoma and Renal Cell Carcinoma
Brief Title: Low-dose Interleukin-2 and Pembrolizumab in Melanoma and Renal Cell Cancer
Acronym: UVA-AM-002
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding was withdrawn
Sponsor: William Grosh, MD (Other)
Responsible Party: Sponsor-Investigator, William Grosh, MD, Associate Professor of Medicine, University of Virginia
Organization: University of Virginia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18537
Record Dates: First submitted 2017-03-23; First posted 2017-04-13 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Renal Cell; Melanoma
Keywords: pembrolizumab; IL-2; interleukin-2; MK-3475
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — pembrolizumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Level 1 (Experimental): Pembrolizumab (200 mg) administered intravenously (day 2 of cycle 1; day 1 of cycles 2 and beyond); Low dose-interleukin 2 (LD-IL2) 12 MIU/m2 administered subcutaneously (days 1-5 and 8-12 of each cycle); each cycle is 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Interleukin-2
- Level -1 (Experimental): Pembrolizumab (200 mg) administered intravenously (day 2 of cycle 1; day 1 of cycles 2 and beyond); Low dose-interleukin 2 (LD-IL2) 5 MIU/m2 administered subcutaneously (days 1-5 and 8-12 of each cycle); each cycle is 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Interleukin-2

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab solution
  Other Names: MK-3475; KEYTRUDA
Drug: Interleukin-2 — Interleukin-2 solution
  Other Names: IL-2

SUMMARY:
This study will evaluate the safety and disease control rate of the combination of pembrolizumab plus low-dose interleukin-2 in patients who have either advanced melanoma or renal cell cancer.

ELIGIBILITY:
Main Inclusion Criteria

* Stage IV or unresectable stage III malignant melanoma or renal cell carcinoma.
* Melanoma

  * Patients must have failed anti-PD-1/PD-L1 antibody therapy.
  * Patients must have failed ipilimumab or be intolerant of ipilimumab and therefore unable to receive ipilimumab.
  * Patients may, but are not obligated, to have failed high- dose IL2.
  * BRAF status must be known or unable to be performed. If the melanoma expresses a BRAF mutation of V600E, V600K, or V600R patient must have received and progressed through a BRAF inhibitor or have failed that therapy due to toxicity.
* Renal Cell Carcinoma

  * Patients must have failed anti-PD-1/PD-L1 antibody therapy.
  * Patients must have failed a VEGF pathway inhibitor and a second tyrosine kinase inhibitor.
  * Patients may, but are not obligated, to have failed high- dose IL2.
* Measurable disease based upon RECIST 1.1.
* Subjects with brain metastases will be eligible if the following are true:
* Subjects with ≤ 3 brain metastases

  * All metastases are ≤ 3 cm
  * All metastases have been treated and are asymptomatic
  * Steroids are not required for management of the brain metastases
  * All metastases have been stable for 1 month following treatment
* Subjects with > 3 brain metastases

  * All metastases are ≤ 3 cm
  * All metastases have been treated and are asymptomatic
  * Steroids are not required for management of the brain metastases
  * All metastases have been stable for 6 months following treatment
* Performance status: ECOG 0-1.
* Adequate organ function.
* Ability to provide informed consent.

Main Exclusion Criteria:

* Pregnancy
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of primary or secondary immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 3 weeks prior to the first dose of trial treatment. Replacement doses of steroids are permitted.
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Known additional malignancies (exceptions DCIS or LCIS, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).
* Prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 3 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Known carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years. Patients may be eligible if they have the following autoimmune diseases: thyroiditis or hypothyroidism, mild arthritis, diabetes, resolved hypophysitis, ulcerative colitis after total abdominal colectomy.
* Active infection requiring systemic therapy.
* Known psychiatric or substance abuse disorders.
* Known history of Human Immunodeficiency Virus (HIV).
* Known active Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Severe chronic pulmonary disease.
* Congestive heart failure, angina, or symptomatic cardiac arrhythmia or is classified according to the New York Heart Association classification as having Class III or IV heart disease.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Safety: adverse event profile | up to 90 days post-treatment
  Obtain preliminary data on the safety of LD-IL2 with pembrolizumab
Disease control rate: melanoma | baseline and every 9 weeks (up to week 104)
  Estimate the disease control rate (CR+PR+SD by RECIST 1.1) among candidate patients with metastatic melanoma treated with pembrolizumab and LD-IL2 and to determine whether disease control is significantly improved. SD for 6 months or more will be considered SD for the purpose of this assessment.
Disease control rate: renal cell cancer | baseline and every 9 weeks (up to week 104)
  Estimate the disease control rate (CR+PR+SD by RECIST 1.1) among patients with metastatic renal cell cancer treated with pembrolizumab and LD-IL2 and to determine whether disease control is significantly improved. SD for 6 months or more will be considered SD for the purpose of this assessment.

SECONDARY OUTCOMES:
Progression free survival: metastatic melanoma | From first response (SD/PR/CR) to time of recurrence/progression or death from any cause, whichever occurs first, assessed for an estimated total of 120 months.
  Estimate progression-free survival defined as the duration of time from first response (SD/PR/CR) to time of recurrence/progression or death from any cause, whichever occurs first
Progression free survival: renal cell cancer | From first response (SD/PR/CR) to time of recurrence/progression or death from any cause, whichever occurs first, assessed for an estimated total of 120 months.
  Estimate progression-free survival defined as the duration of time from first response (SD/PR/CR) to time of recurrence/progression or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: William W Grosh, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No